CLINICAL TRIAL: NCT02867969
Title: Slowing Down Disease Progression in Premanifest SCA: a Piloting Interventional Exergame Trial
Acronym: SlowSCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SlowSCA
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Spinocerebellar Ataxia
Keywords: Spinocerebellar ataxia; Exergaming; Neurodegenerative diseases; Rare disease; Motor exercises; Premanifest stage; Training
MeSH Terms: conditions — Spinocerebellar Ataxias; Neurodegenerative Diseases; Rare Diseases | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motor training (Other): The motor training comprise of demanding coordinative exercises based on commercially available developed by Microsoft Game Console (XBOX Kinect™) exergames that specifically target ataxia dysfunctions.
  Interventions: Other: Motor training

INTERVENTIONS:
Other: Motor training — The motor training will comprise of demanding coordinative exercises based on commercially available developed by Microsoft Game Console (XBOX Kinect™) exergames that specifically target ataxia dysfunctions.
  Other Names: Exergaming

SUMMARY:
This is a piloting study using continuous motor training provided via whole body-controlled video games (exergames) to establish proof-of-concept evidence that such training leads to motor and neural changes in pre-manifest subjects with spinocerebellar ataxias (SCA).

DETAILED DESCRIPTION:
In many neurodegenerative diseases, including spinocerebellar ataxias (SCA), large populations of neurons are already lost and compensatory resources exhausted at time of clinical diagnosis. This calls for early intervention strategies aiming to slow down disease progression already at the premanifest stage of the disease. Here we propose the world-first interventional study aiming to delay onset in a rare genetic neurodegenerative disease. Specifically, we propose a piloting study using continuous motor training provided via whole body-controlled video games (exergames) to establish proof-of-concept evidence that such training leads to motor and neural changes in pre-manifest SCA subjects. The subclinical effects will be unravelled within an intraindividual control study design by elaborated quantitative Video Management System (VICON®)-based movement analysis and structural and functional 3 Tesla (T) magnetic resonance imaging. This will provide unique insights in underlying motor and neural networks and compensatory strategies. If successful, this piloting trial will provide the basis for a rigorous international multi-center large-scale study in a larger SCA population. Moreover, it will stimulate complementary tandem projects on effects of motor training on neural functioning and molecular pathways in premanifest SCA mouse models.

ELIGIBILITY:
Inclusion Criteria:

* adult persons (age 18-80 years) who (i) are a blood-related relative of an index subject with a known SCA 1,2,3 or 6 mutation and who (ii) have a score value of <8 points on the Scale for the Assessment and Rating of Ataxia (SARA)
* full capacity to consent to study participation after extensive information (fully Informed Consent)

Exclusion Criteria:

* Cognitive deficits which prevent full comprehension of the study requirements and/or training requirements
* Comorbid diseases that place severe constraints on a continous training with whole-body controlled exergames (e.g. severe visual or hearing deficits; severe paresis; severe movement disorders other than ataxia)
* Comorbid neurologic disease other than ataxia (e.g. prior stroke or brain trauma)
* Pregnant or breast-feeding persons
* Lack of capacity for full informed consent according to established psychiatric criteria for full informed consent

Magnetic Resonance Imaging (MRI) exclusion criteria:

* cardiac pacemakers
* artificial heart valves
* metal prostheses
* implanted magnetic metal parts (screws, plates and similar devices)
* intrauterine devices (for instance, for contraceptive purposes)
* shrapnel parts and other metal pieces
* non-removable braces and metal dentures
* non-removable acupuncture needles
* insulin pumps and infusion ports
* tattoos, eye shadow and other metal-containing make-up
* The subject has decreased sensitivity to temperature and / or decreased tolerance towards elevated body temperatures or warming of body parts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Gait score | Day 43
  Decrease in a quantitative composite gait score consisting of body sway and gait variability in walking challenge conditions (mattress), assessed by VICON-based motion tracking

SECONDARY OUTCOMES:
Brain networks captured | Day 43
  Changes in brain networks captured by specific neuroimaging focussing on brain grey matter volume (VBM), brain fibre tracking (DTI) and functional connectivity of the cerebellum with other brain regions (resting-state connectivity)
Quantitative movement parameters | Day 43
  Set of quantitative movement parameters for complex whole-body movements (gait, stand, fast sequences of goal-directed stepping movements) (VICON-based motion tracking).
Ataxia severity | Day 43
  Clinical ataxia severity according to the Scale for the Assessment and Rating of Ataxia (SARA)
Daily activity | Day 43
  Objectively measured level of daily activity in subjects' real-world settings (body-worn motions sensors; ActivePal®)
Brain-derived neurotrophic factor | Day 43
  Increase of serum brain-derived neurotrophic factor (BDNF)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No